CLINICAL TRIAL: NCT03656406
Title: Effect of Lateral Positioning on Bronchial Cuff Pressure of Left-sided Double-lumen Endotracheal Tube During Thoracic Surgery: a Prospective Observational Study
Brief Title: Effect of Lateral Positioning on Bronchial Cuff Pressure of Left-sided Double-lumen Endotracheal Tube During Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: Daegu Catholic University Medical Center (Other)
Collaborators: Research Institute of Medical Science, Daegu Catholic University (Unknown)
Responsible Party: Principal Investigator, Sung Hye Byun, Assistant Professor, Daegu Catholic University Medical Center
Other Study IDs: CR-18-111
Record Dates: First submitted 2018-08-30; First posted 2018-09-04 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Lung Cancer; Pneumothorax
Keywords: Double-lumen endotracheal tube; Cuff pressure
MeSH Terms: conditions — Lung Neoplasms; Pneumothorax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Behavioral: Lateral decubitus positioning — After the DLT intubation, the patient is placed in lateral decubitus position
Device: Cuff-manometer — The pressure of the bronchial cuff should be measured with cuff-manometer in supine position, and then measurement should be repeated after lateral positioning.

SUMMARY:
The investigators evaluate the effect of postural change on the bronchial cuff pressure (BCP) of double-lumen endotracheal tube (DLT) in patients undergoing thoracic surgery, by observing the pressure of the bronchial cuff before and after lateral decubitus positioning.

DETAILED DESCRIPTION:
It is essential to maintain proper cuff pressure in the endotracheal tube (ETT) when placing the ETT in the trachea in patients undergoing general anesthesia. Most of the literature recommend maintaining a pressure of 20-30 cmH2O to prevent cuff-related complications such as micro-aspiration or airway trauma. Proper pressure is also important for DLTs used in thoracic surgery. Furthermore, the cuff pressure of the ETT can change during the patient's positional changes. All things considered, we hypothesized that the change from supine to lateral decubitus position, which is essential for thoracic surgery would affect the BCP of the DLT.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status 1 or 2
2. Elective lung surgery requiring lateral decubitus positioning and one-lung ventilation using left-sided DLT

Exclusion Criteria:

1. Patients requiring a right-sided DLT.
2. Patients with an intraluminal lesion in the left mainstem bronchus (LMB).
3. Patients with an anatomical problem in the tracheobronchial tree.
4. Patients with impaired lung such as chronic obstructive pulmonary disease.
5. Patients who refused to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-70 years with an American Society of Anesthesiologists (ASA) physical status 1 or 2, who are scheduled to undergo elective lung surgery requiring lateral decubitus positioning and one-lung ventilation (OLV) using left-sided DLT
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Change of the maximum bronchial cuff pressure (BCP) which does not exceed 40 cmH2O with no air leak from supine to lateral decubitus position | 1. In supine position, 2 minutes after the completion of confirming the double-lumen endotracheal tube (DLT) position via fiberoptic bronchoscope (FOB) 2. In lateral position, 2 minutes after the completion of confirming the DLT position via FOB
  A cuff-manometer will be connected to the valve of the pilot balloon of bronchial cuff via a three-way stopcock. And then, the BCP will be assessed, while inflating the cuff with air in 0.5 ml increments from 0 to 3.0 ml. If the BCP exceeds 40 cmH2O during expansion by increasing 0.5 ml from 0 to 3.0 ml, we will stop inflating the bronchial cuff with air and record the bronchial cuff volume (BCV) and BCP up to the last numerical value. During the pressure measurement, air leak or seal around the bronchial cuff will be assessed at each time point when inflating the cuff in 0.5 ml increments.

SECONDARY OUTCOMES:
The incidence of the patients whose maximum BCP exceed 40 cmH2O after lateral positioning | 1. In supine position, 2 minutes after the completion of confirming the DLT position via FOB 2. In lateral position, 2 minutes after the completion of confirming the DLT position via FOB
The minimum BCV that is the smallest bronchial cuff volume without air leakage | 1. In supine position, 2 minutes after the completion of confirming the DLT position via FOB 2. In lateral position, 2 minutes after the completion of confirming the DLT position via FOB

CONTACTS AND LOCATIONS:
Locations (1):
- Sung-Hye Byun, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu CY, Yeh YC, Wang MC, Lai CH, Fan SZ. Changes in endotracheal tube cuff pressure during laparoscopic surgery in head-up or head-down position. BMC Anesthesiol. 2014 Aug 31;14:75. doi: 10.1186/1471-2253-14-75. eCollection 2014. PMID 25210501
- [Background] Athiraman U, Gupta R, Singh G. Endotracheal cuff pressure changes with change in position in neurosurgical patients. Int J Crit Illn Inj Sci. 2015 Oct-Dec;5(4):237-41. doi: 10.4103/2229-5151.170841. PMID 26807392
- [Background] Araki K, Nomura R, Urushibara R, Yoshikawa Y, Hatano Y. Bronchial cuff pressure change caused by left-sided double-lumen endobronchial tube displacement. Can J Anaesth. 2000 Aug;47(8):775-9. doi: 10.1007/BF03019480. PMID 10958094
- [Derived] Kim E, Kim IY, Byun SH. Effect of lateral positioning on the bronchial cuff pressure of a left-sided double-lumen endotracheal tube during thoracic surgery: study protocol for a prospective observational study. BMJ Open. 2019 Mar 30;9(3):e026606. doi: 10.1136/bmjopen-2018-026606. PMID 30928955